CLINICAL TRIAL: NCT05476757
Title: Safety, Virological and Immunological Assessment of the Controlled Dengue Human Infection Model in Thailand
Brief Title: Safety, Virological and Immunological Assessment of Live Attenuated Dengue Serotype 2 rDEN2delta30-7169.
Acronym: DHIT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 022/2565(IRB1)
Record Dates: First submitted 2022-07-11; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Dengue
Keywords: Controlled Human Infection Model; Flavivirus naïve
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: 5 flavivirus naïve participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flavivirus naïve (Experimental)
  Interventions: Biological: rDEN2Δ30-7169

INTERVENTIONS:
Biological: rDEN2Δ30-7169 — rDEN2Δ30-7169 will be inoculated at Study Day 0. After 6 months of the inoculation, the participants will be vaccinated with Dengvaxia® until completion of 3 doses with 6-month interval between each dose.

SUMMARY:
Dengue viral infection and dengue hemorrhagic fever (DHF) are important emerging health problems worldwide. Several candidate dengue vaccines are currently in different stages of development but CYD is the only licensed vaccine currently available. Although this vaccine can induce neutralizing antibodies against all four DENV serotypes, the vaccine showed enhanced hospitalization in recipients who were dengue-naïve before vaccination. The long-term safety assessment of the vaccine in endemic regions demonstrated that the risk of hospitalization in year 3 of vaccination was higher in the vaccine group especially among recipients under 9 years of age with a relative risk of 1.58 [95% CI, 0.83 to 3.02].

Surrogate animal models are not good models to see whether the vaccine or therapeutic is able to be tested in clinical trials since animals do not develop symptoms of infection as in humans. The ADE phenomenon and the lack of known correlates of protection in animal models are still the major problems and challenges in the development of an effective dengue vaccine and make it difficult to identify candidate vaccines. The efficacy and safety situation of CYD also highlights the requirement of verification of candidate vaccines before performing clinical trials with a large number of participants.

The controlled human infection model, therefore, has been proposed to pre-evaluate candidate vaccines before moving into larger clinical trials. It has been previously used for several infectious diseases i.e., malaria, norovirus, influenza, cholera, Campylobacter, and Shigella, to accelerate vaccine or therapeutic development. For dengue, two controlled dengue human infection models (DHIM) have been established for vaccine testing and evaluation of therapeutics in a dengue naïve population in the USA. Although it has been proved useful for studies of dengue in naïve individuals, it is necessary to set up DHIM in endemic regions like Thailand as more than 90% of the population has been previously exposed to the virus and, importantly, host immune status prior to the introduction of viruses can influence clinical outcomes and vaccine efficacy. It will also be very challenging in terms of safety concerns since having pre-existing immune responses to natural DENV infection is a risk factor for severe dengue. The establishment of DHIM will not only allow a small-scale demonstration for safety and efficacy of vaccines or therapeutics which can appropriately guide the design of phase III to be more cost-effective but it will also allow the investigation of immune correlates of protection and determination of factors correlated with disease protection and pathogenesis as clinical endpoints can be closely followed up in all participants.

Safety, Virological and Immunological Assessment of the Controlled Dengue Human Infection Model in Thailand (DHIT) is proposed to challenge the live attenuated dengue virus serotype 2, rDEN2Δ30-7169, in 5 flavivirus naïve participants recruited from Bangkok, Thailand, and aims to assess the safety, viremia, NS1 antigenemia profile, and immunogenicity of the challenge virus in the volunteers.

In addition, this DHIT project will vaccinated all 5 participants with Dengvaxia® after inoculation with the challenge virus to reduce the risk of severe disease of dengue in the future. Blood collection will be obtained after each vaccination to assess virological and immunological profiles. Active and passive surveillance will be set up to monitor for dengue infection after vaccination. The overall study period from administration of live attenuated virus until last follow-up visit is 38 months.

ELIGIBILITY:
Inclusion Criteria:

1. Thai healthy volunteers, aged between 18 to 30 years old and weight is greater than or equal to 45 kg and have Thai language literacy.
2. Don't have any history of previous dengue, zika or Japanese encephalitis virus infection
3. Have not given blood donation in the past 3 months
4. Education: higher than high school
5. Display flavivirus immunity profile defined by the standard PRNT 50% (PRNT50) as follows: flavivirus naïve is defined as the PRNT50 titer against

   * DENV1 < 1:5
   * DENV2 < 1:5
   * DENV3 < 1:5
   * DENV4 < 1:5
   * ZIKV < 1:5
   * JEV < 1:5
6. Willingness to participate in the study as evidenced by signing the informed consent document.
7. Female participants of childbearing potential should be agreed to either abstinence or use at least one primary form of contraception from the time of screening for rDEN2Δ30-7169 administration until 1 month after complete course of Dengvaxia® vaccination (Study Day 568).

Exclusion Criteria:

1. For female participants: Currently pregnant, as determined by positive β-human choriogonadotropin (HCG) test or breast-feeding, and given birth or abortion within 6 months.
2. History of previous acute undifferentiated febrile illness leading to hospitalization in the past 3 months
3. Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperate with the requirements of the study protocol.
4. Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history.
5. History of a severe allergic reaction or anaphylaxis
6. Severe asthma (emergency room visit or hospitalization within the last 6 months).
7. Any known immunodeficiency syndrome.
8. Having any pre-existing medical conditions consist of thrombocytopenia, autoimmune disease and cancer based on history, physical examination, and/or laboratory studies.
9. Current use of anticoagulant medications (this includes anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
10. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. An immunosuppressive dose of corticosteroids is defined as ≥ 10 mg of a prednisone equivalent per day for ≥ 14 days.
11. Asplenia
12. Receipt of any vaccine within 28 days or a killed vaccine within 14 days prior to receive virus administration, or anticipated receipt of any vaccine during the 28 days following rDEN2∆30-7169 administration.
13. Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following rDEN2∆30-7169 administration.
14. Previous receipt of a flavivirus vaccine (licensed or experimental).
15. Screening laboratory values of Grade 1 or above (as defined in this protocol) for ANC (<750 /mm3), Platelet (<100,000 /mm3), PT (> 1.25 x ULN), APTT (> 1.66 x ULN), ALT (>2.5 x ULN) and serum creatinine (> 1.3 x ULN OR Increase to >1.3 x participant's baseline)
16. Body temperature higher than 37.5 °C
17. HIV infection, as indicated by anti-HIV screening assays.
18. Hepatitis C virus (HCV) infection, as indicated by anti-HCV screening assays.
19. Hepatitis B virus (HBV) infection, as indicated by hepatitis B surface antigen (HBsAg) and/or anti-HBc screening.
20. Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The safety of rDEN2Δ30-7169 in flavivirus naïve participants | 21 Days
  Occurrence of local and general adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
The frequency of viremia following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Proportion of number of volunteer with detectable virus genome assessed by nested RT-PCR, real time RT-PCR and virus culture after administration of DENV2Δ30-7169
The quantity of viral genome following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  The quantity of viral genome (copies/mL) assessed by nested RT-PCR, real time RT-PCR and virus culture after administration of DENV2Δ30-7169
The duration of viremia following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Days of detectable virus genome assessed by nested RT-PCR, real time RT-PCR and virus culture after administration of DENV2Δ30-7169
The frequency of viremia following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Proportion of number of volunteer with detectable infectious activity assessed by nested RT-PCR, real time RT-PCR and virus culture after administration of DENV2Δ30-7169
The quantity of infectious activity following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  The quantity of infectious activity (FFU/mL) assessed by nested RT-PCR, real time RT-PCR and virus culture after administration of DENV2Δ30-7169
The duration of infectious activity following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Days of detectable infectious activity assessed by nested RT-PCR, real time RT-PCR and virus culture after administration of DENV2Δ30-7169
The frequency of NS1 antigenemia following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Proportion of number of volunteer with detectable NS1 antigen after administration of DENV2Δ30-7169
The quantity of NS1 antigenemia following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  The quantity of NS1 antigenemia (ng/mL) after administration of DENV2Δ30-7169
The duration of NS1 antigenemia following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Days of detectable NS1 antigen after administration of DENV2Δ30-7169
The immunogenicity of rDEN2Δ30-7169 in Thai flavivirus naïve participants | 180 Days
  Levels of neutralizing antibodies (NT50) as measured by PRNT to dengue virus after administration with rDEN2Δ30-7169
Measurement of levels of anti-dengue virion-IgM/IgG antibodies following administration with rDEN2Δ30-7169 in flavivirus naïve participants | 180 Days
  Levels of anti-dengue virion-IgM/IgG antibodies (titer) as measured by ELISA following administration with rDEN2Δ30-7169 in flavivirus naïve participants

OTHER OUTCOMES:
The cellular immune responses including dengue virus specific B cells and NS3 peptides specific T cells to all four DENV serotypes following administration of rDEN2Δ30-7169 in Thai flavivirus naïve participants | Study Day 0-60
  The frequency of dengue virus specific B cells and NS3 peptides specific T cells (percentage of cells/total lymphocytes) to all four DENV serotypes following administration of rDEN2Δ30-7169 in Thai flavivirus naïve participants
To measure anti-dengue virion-IgM/IgG antibodies following vaccination with Dengvaxia® | Study Day 194-1140
  Levels of anti-dengue virion-IgM/IgG antibodies (titer) as measured by ELISA following vaccination with Dengvaxia®
The immunogenicity following vaccination with Dengvaxia® | Study Day 194-1140
  Levels of neutralizing antibodies (NT50) as measured by PRNT to dengue virus following vaccination with Dengvaxia®
The frequency of viremia in oral fluid specimens following administration with rDEN2Δ30-7169 | Study Day 0-600
  Proportion of number of volunteer with viremia as assessed by RT-PCR oral fluid specimens following administration with rDEN2Δ30-7169 and vaccination with Dengvaxia®
The quantity of viremia in oral fluid specimens following administration with rDEN2Δ30-7169 | Study Day 0-600
  The quantity of viremia (copies/mL) as assessed by RT-PCR oral fluid specimens following administration with rDEN2Δ30-7169 and vaccination with Dengvaxia®
The duration (days) of viremia in oral fluid specimens following administration with rDEN2Δ30-7169 | Study Day 0-600
  Days of viremia as assessed by RT-PCR oral fluid specimens following administration with rDEN2Δ30-7169 and vaccination with Dengvaxia®
Anti-NS1 antibodies and anti-dengue IgM, IgG, IgG1, IgA antibodies levels in oral fluid specimens following administration with rDEN2Δ30-7169 and vaccination with Dengvaxia® in Thai flavivirus naïve participants | Study Day 0-600
  Levels of anti-NS1 antibodies and anti-dengue IgM, IgG, IgG1, IgA antibodies (unit) as measured by ELISA in oral fluid specimens following administration with rDEN2Δ30-7169 and vaccination with Dengvaxia® in Thai flavivirus naïve participants

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand